CLINICAL TRIAL: NCT06973200
Title: Epidemiological Profile of Schistosomiasis and Soil-transmitted Helminth Infections Among Schoolchildren in Banfora Municipality, Burkina Faso: a Pilot Study
Brief Title: Burden of Schistosomiasis and Soil-transmitted Helminth Infections in Schoolchildren in Banfora, Burkina Faso
Acronym: NTDs_SAC
Status: Completed | Type: Observational
Sponsor: Centre MURAZ/Institut National de Santé Publique (Other Government)
Collaborators: Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government); University of Ghana (Other)
Responsible Party: Sponsor
Other Study IDs: INSP_CM_08_2024; ACE02-WACCBIP (Other Grant/Funding Number: World Bank/WACCBIP, University of Ghana)
Record Dates: First submitted 2025-02-03; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-01

CONDITIONS: Schistosomiasis in Children; Soil Transmitted Helminth (STH) Infections; Malaria Infection; Anaemia; Malnutrition in Children
Keywords: Epidemiology of schistosomiasis and STH infections; Efficacy and safety of dihydroartemisinin-piperaquine
MeSH Terms: conditions — Infections; Anemia; Child Nutrition Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, stool, and urines samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | US Export: No

INTERVENTIONS:
Combination Product: Dihydroartemisin-piperaquine — All children with S. mansoni and/or S. haematobium infections at enrolment will then be treated with dihydroartemisinin-piperaquine (DP) and followed up on days 1, 2, 3, 4, 28, and 42 to assess the efficacy and safety of DP.

SUMMARY:
A cross-sectional study will be conducted among 300 schoolchildren in the Banfora region, including 120 in urban and 180 in rural areas, to assess the prevalence of schistosomiasis and soil-transmitted helminth infections. All children with S. mansoni and/or S. haematobium infections at enrolment will then be treated with dihydroartemisinin-piperaquine (DP) and followed up on days 1, 2, 3, 4, 28, and 42 to assess the efficacy and safety of DP. At the end of the study, all children (infected and uninfected) will receive praziquantel and albendazole according to national recommendations.

DETAILED DESCRIPTION:
At enrolment, pre-tested structured questionnaire will be administered to each enrolled child and his/her parent or legal guardian to collect socio-demographic data (age, sex, class), exposure factors to schistosomiasis and soil-transmitted helminth infections (eating and drinking habits, wearing of shoes, use of latrines and contact with water) and disease history. In addition, the child's clinical data (body temperature, weight and height) will be collected. Axillary temperature is measured with an electronic thermometer. Weight and height are measured using a mechanical scale and a height gauge with an accuracy of 0.1 cm and 0.1 kg, respectively, according to standard procedures.

A venous blood sample (4 mL) will then be taken to test for malaria and to measure haemoglobin concentration. The remaining blood sample will be stored for future study. Children with confirmed malaria infection or anaemia will be treated with dihydroartemisinin-piperaquine (DP) or iron folic acid according to national recommendations. In addition, each participant will receive two pre-labeled (identification code and date) sterile plastic containers to collect stool and urine samples. The stool samples will be used to diagnose S. mansoni infection and soil-transmitted helminth infections, while the urine samples will be used to detect circulating S. mansoni antigens and S. haematobium eggs. The urine samples will be collected on the day of enrolment, while the stool containers will be collected the following morning (each child will be instructed to place part of their stool sample in the container). Part of the biological samples will be processed in the laboratory of the Banfora Urban Medical Centre. The remaining biological samples will then be stored in the same laboratory before being transported in refrigerated containers to the Parasitology-Mycology Laboratory of the Centre MURAZ, where they will be archived for ten years.

Upon enrolment, only children infected with S. mansoni and/or S. haematobium will be treated with DP and followed up on days 1, 2, 3, 4, 28, and 42 to assess the efficacy and safety of DP. Project nurses will administer all doses of DP, and participants will be monitored for 30 minutes. Any participant who vomits during the first 30 minutes will be given a replacement dose. Participants with repeated vomiting will be excluded from the study and managed according to national guidelines. However, at the end of the study, all schoolchildren will be treated with PZQ (40 mg/kg) and albendazole (400 mg) according to national guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Age between 5 and 15 years;
* Resident in Banfora town for at least 6 months before the start of the study;
* Assent of the child (over 12 years of age);
* Informed consent from the child's parent or legal guardian.

Exclusion Criteria:

* Use of praziquantel and albendazole in the past 6 months;
* Use of Artemisinin-based combination therapies (ACTs) in the 3 weeks before study start-up;
* Known allergy to DP;
* Current episode of diarrhoea;
* Inability to provide stool and urine samples;
* Child absent on the day of the survey.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Schoolchildren from the five selected primary schools in the Banfora community will be included in the study.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2024-12-21 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
Prevalence of schistosomiasis and soil-transmitted helminth (STH) infections | January 2025
  Porportion of children infected by schistosomes and soil-transmitted helminths. S. mansoni and STHs will be screened using the Kato Katz method while S. haematobium will be detected using the urine filtration method.
Intensity of S. mansoni and soil-transmitted helminth (STH) infections | January 2025
  The intensity of S. mansoni and STH infections will be determined using the Kato-Katz method and expressed as the number of eggs per gram of feces.
Intensity of S. haematobium infection | January 2025
  The intensity of S. haematobium infection will be determined using urine filtration method and expressed as the number of eggs per 10 mL of urine.
Risk factors associated with schistosomiasis and soil-transmitted helminth infections | January 2025
  Potential predictors of schistosomiasis and soil-transmitted helminth infections, such as study participants' socio-demographic data, WASH conditions, and exposure to water bodies, will be collected using a structured questionnaire.
  Multivariable logistic regression will be used to explore predictors significantly associated with the prevalence of schistosomiasis and soil-transmitted helminth infections.

SECONDARY OUTCOMES:
Cure rate (CR) | 4 weeks and 6 weeks after starting DP treatment
  The CR is defined as the proportion of egg-positive children at baseline, who become egg-negative after DP treatment in all collected stool or urine samples.
Eggs reduction rate (ERR) | 4 weeks and 6 weeks after DP treatment
  The ERR (defined as the proportional reduction in the mean eggs per gram of faeces (S. mansoni) or per ml of urine (S. haematobium) post-treatment versus pre-treatment)), as assessed by microscopy.
Drug-related adverse events | First 4 weeks after DP treatment
  The number of participants with drug-related adverse events or serious adverse events
Prevalence of malaria among schoolchildren | January 2025
  Proportion of children infected with malaria parasites as determined by microscopy and rapid diagnostic test
Risk factors of malaria among schoolchildren | January 2025
  Potential predictors of malaria including study participants' socio-demographic data and exposure to malaria will be collected using a structured questionnaire. Then predictors significantly associated with the prevalence of malaria will be explored using a multivariable logistic regression.
Prevalence of anaemia among schoolchildren | January 2025
  Proportion of children with anaemia will determined and anaemia will be defined on the basis of haemoglobin concentration according to (WHO, 2011). Haemoglobin concentration will be measured using a Hemocue photometer from a venous blood sample.
Risk factors of anaemia among schoolchildren | January 2025
  Key predictors of anaemia, including study participants' socio-demographic data, malaria infection, and helminth infection (i.e, schistosomiasis and STHs infection), will be collected using a structured questionnaire. Then predictors significantly associated with the prevalence of anaemia will be identified using a multivariable logistic regression.

CONTACTS AND LOCATIONS:
Overall Officials: Mamoudou Cissé, MD, MSc, PhD, Principal Investigator — Centre MURAZ/Université Nazi BONI
Locations (1):
- Banfora, Banfora, Comoé, Burkina Faso